CLINICAL TRIAL: NCT06080997
Title: Patients' Expectations Before, and Their Experiences After Spinal Surgery, Regarding Pain, Rehabilitation and Quality of Life
Brief Title: Patients' Expectations Before Spinal Surgery
Status: Recruiting | Type: Observational
Sponsor: Zealand University Hospital (Other)
Responsible Party: Principal Investigator, Josephine Zachodnik, PhD student, Zealand University Hospital
Other Study IDs: EXP - jzc - 2023
Record Dates: First submitted 2023-10-06; First posted 2023-10-12 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Expectations; Surgery; Pain; Quality of Life
Keywords: Expectations; Pain; Rehabilitation; Quality of life
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Spinal surgery: No intervention will take place Recruiting autumn 2023 until autumn 2024. All patients at Zealand University Hospital, who meet the inclusion criteria, undergoing spinal surgery during 1 year, will be invited to participate in the quantitative part of the study.
  We estimate that 300 patients will be eligible for the quantitative part. For the qualitative part, we will include 10 - 15 patients undergoing spinal surgery.

SUMMARY:
With this study the investigators want to perform a prospective observational cohort study at Zealand University Hospital, Koege, Denmark.

The purpose of this study is twofold:

1. to investigate how expectations predict patients' pain, rehabilitation and quality of life after spinal surgery.
2. to explore the patients' expectations before, and their experiences after, spinal surgery regarding pain, rehabilitation and quality of life.

DETAILED DESCRIPTION:
Background Surgery can be an overwhelming and often life-changing experience for patients. To mitigate this experience a patient-centered approach can be beneficial. Patient-centered care is defined as providing care that is "respectful of and responsive to individual patient preferences, needs and values, and which ensures that patient values guide all clinical decisions". Patient-centeredness should be considered in discussions about the value of surgical treatment for the patient and the expectations regarding the process of postoperative rehabilitation, especially considering the patient's definition of a successful outcome. The meaning of rehabilitation may vary between stakeholders involved in surgery, including patients, surgeons, anaesthetists, nurses, and hospital administrators. Studies addressing strategies to improve rehabilitation, such as minimally invasive surgery and enhanced recovery pathways, commonly focus on measures such as complication rates, gastrointestinal activity, physical function, and duration of hospital stay. These parameters are mostly relevant to clinicians and administrators, but they do not reflect the complexity of the rehabilitation process or include the patient's perspective and expectations.

In musculoskeletal practice, patients' expectations have been reported as a valuable predictor for treatment outcomes in patients with acute and chronic pain. Patients with higher expectations regarding the treatment report better outcomes than those with lower expectations. Previous studies have investigated the relationship between expectations and postoperative satisfaction in patients undergoing spinal surgery, and some evidence suggests patients' expectations also impact rehabilitation after surgery.

Patients undergoing spinal surgery usually suffer from moderate to severe pain during the perioperative and postoperative period, which is associated with developing persistent pain 8 and compromises patients' quality of life.

Lumbar disc herniation is one of the most common musculoskeletal diseases which, in some cases, can compromise patients' quality of life, and the most common operations performed on the spine. A previous study has shown that persistent pain after surgery for lumbar disc herniation is negatively associated with psychological and physical well-being, and the overall quality of life is decreased.

This study hypothesize that interviewing patients in a semi-structured manner would give unique perspectives on what is important to patients, as opposed to what is important to researchers. Further, the study hypothesize that patients' preoperative expectations for spinal surgery can affect postoperative rehabilitation. Gaining an in-depth understanding of the process of recovery from the patient´s perspective can, ultimately, guide patient-centered care and future research.

ELIGIBILITY:
Inclusion Criteria:

Patients undergoing elective spinal surgery. Patients able to read and understand Danish.

Exclusion Criteria:

Patients with cognitive deficits, such as dementia. Patients with alcohol and drug dependence.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients at Zealand University Hospital, undergoing spinal surgery during 1 year, will be invited to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Expectations | Outcome measure will be assessed and presented 2025
  Expectations measured by Treatment Expectation Questionnaire (TEX Q) pre-operatively and 3 month postoperatively
Patients Expectations | Outcome measure will be assessed and presented 2025
  Expectations measured by a semi-structured interview pre-operatively

SECONDARY OUTCOMES:
Patients pain intensity | Outcome measure will be assessed and presented 2025
  Pain level measured by Verbal Rating Scale (VRS) pre-operatively and 3 month post- operatively
Patients functional level | Outcome measure will be assessed and presented 2025
  Functional level measured by Oswestry Disability Index (ODI) pre-operatively and 3 month post-operatively
Quality of life score | Outcome measure will be assessed and presented 2025
  Quality of life measured by WHO Quality of Life - BREF (WHOQOL-BREF) pre-opertively and 3 month post-operatively

CONTACTS AND LOCATIONS:
Overall Officials: Anja Geisler, Study Director — Zealand University Hospital Koege
Locations (1):
- Zealand University Hospital, Køge, Region Sjælland, Denmark

REFERENCES:
- [Background] Rajabiyazdi F, Alam R, Pal A, Montanez J, Law S, Pecorelli N, Watanabe Y, Chiavegato LD, Falconi M, Hirano S, Mayo NE, Lee L, Feldman LS, Fiore JF Jr. Understanding the Meaning of Recovery to Patients Undergoing Abdominal Surgery. JAMA Surg. 2021 Aug 1;156(8):758-765. doi: 10.1001/jamasurg.2021.1557. PMID 33978692
- [Background] Lee L, Tran T, Mayo NE, Carli F, Feldman LS. What does it really mean to "recover" from an operation? Surgery. 2014 Feb;155(2):211-6. doi: 10.1016/j.surg.2013.10.002. Epub 2013 Oct 12. No abstract available. PMID 24331759
- [Background] Mohamed Mohamed WJ, Joseph L, Canby G, Paungmali A, Sitilertpisan P, Pirunsan U. Are patient expectations associated with treatment outcomes in individuals with chronic low back pain? A systematic review of randomised controlled trials. Int J Clin Pract. 2020 Nov;74(11):e13680. doi: 10.1111/ijcp.13680. Epub 2020 Sep 7. PMID 33166045
- [Background] Krauss P, Sonnleitner C, Reinartz F, Meyer B, Meyer HS. Patient-Reported Expectations, Outcome and Satisfaction in Thoracic and Lumbar Spine Stabilization Surgery: A Prospective Study.Surgeries 2020; 1: 63-76.
- [Background] Werner MU, Mjobo HN, Nielsen PR, Rudin A. Prediction of postoperative pain: a systematic review of predictive experimental pain studies. Anesthesiology. 2010 Jun;112(6):1494-502. doi: 10.1097/ALN.0b013e3181dcd5a0. PMID 20460988
- [Background] Frisaldi E, Shaibani A, Benedetti F. Why We should Assess Patients' Expectations in Clinical Trials. Pain Ther. 2017 Jun;6(1):107-110. doi: 10.1007/s40122-017-0071-8. Epub 2017 May 5. PMID 28477082
- [Background] Gerbershagen HJ, Aduckathil S, van Wijck AJ, Peelen LM, Kalkman CJ, Meissner W. Pain intensity on the first day after surgery: a prospective cohort study comparing 179 surgical procedures. Anesthesiology. 2013 Apr;118(4):934-44. doi: 10.1097/ALN.0b013e31828866b3. PMID 23392233
- [Background] Gulur P, Nelli A. Persistent postoperative pain: mechanisms and modulators. Curr Opin Anaesthesiol. 2019 Oct;32(5):668-673. doi: 10.1097/ACO.0000000000000770. PMID 31343465
- [Background] Papadopoulos T, Abrahim A, Sergelidis D, Bitchava K. Original article Ερευνητική. 2011; 2: 119-23.
- [Background] Heider D, Kitze K, Zieger M, Riedel-Heller SG, Angermeyer MC. Health-related quality of life in patients after lumbar disc surgery: a longitudinal observational study. Qual Life Res. 2007 Nov;16(9):1453-60. doi: 10.1007/s11136-007-9255-8. Epub 2007 Sep 12. PMID 17849238
- [Background] Kong H, West S. WMA DECLARATION OF HELSINKI - ETHICAL PRINCIPLES FOR Scienti c Requirements and Research Protocols. 2013; 29-32.
- [Background] Alberts J, Lowe B, Glahn MA, Petrie K, Laferton J, Nestoriuc Y, Shedden-Mora M. Development of the generic, multidimensional Treatment Expectation Questionnaire (TEX-Q) through systematic literature review, expert surveys and qualitative interviews. BMJ Open. 2020 Aug 20;10(8):e036169. doi: 10.1136/bmjopen-2019-036169. PMID 32819942
- [Background] Graneheim UH, Lundman B. Qualitative content analysis in nursing research: concepts, procedures and measures to achieve trustworthiness. Nurse Educ Today. 2004 Feb;24(2):105-12. doi: 10.1016/j.nedt.2003.10.001. PMID 14769454

DOCUMENTS (1):
  • Study Protocol (2023-05-09): https://cdn.clinicaltrials.gov/large-docs/97/NCT06080997/Prot_000.pdf